CLINICAL TRIAL: NCT05585723
Title: French Language Validation of Questionnaires for the Evaluation of Problematic Screen Use.
Acronym: VALSCREEN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A01943-40
Record Dates: First submitted 2022-10-10; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Smartphone Addiction
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- students at the university
  Interventions: Behavioral: Questionnaires completion
- teenagers
  Interventions: Behavioral: Questionnaires completion
- parents of teenagers
  Interventions: Behavioral: Questionnaires completion

INTERVENTIONS:
Behavioral: Questionnaires completion — Prospective, qualitative, observational, single-center study. 1) Two independent translations of the original questionnaires into French, 2) Back-translation of the consensus version into English by a professional bilingual translator 3) We will submit this final version to two opinion leaders in France. 4) Evaluation of the clarity, comprehension and acceptability of the translation of the questionnaire.

SUMMARY:
The main objective of this research is to linguistically validate the Smartphone Addiction Scale, Nomophobia Questionnaire, The Problematic Use of Mobile Phones scale, Smartphone Addiction Proneness Scale, Digital Addiction Scale for Children, Gaming Motivation Scale and Problematic Media Use Measure in French so that they are conceptually equivalent to their original version.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the SAS, NMP-Q, SAPS questionnaires
* University students over 18 years of age Inclusion criteria for the GAMS questionnaire
* University students over 18 years of age
* Video game players (at least one video game session in the past two weeks) Inclusion criteria for the PUMP and DASC questionnaires
* Adolescents (12-17 years old) Inclusion criteria for the PMUM-SF questionnaire
* Parents of adolescents (this can be parents of adolescents who answered the previous questions)
* Adolescents must have access to at least one screen: smartphone, computer, television, etc (even that of a parent)

Exclusion Criteria:

* Difficulties in understanding the French language
* Cognitive disorders
* Subject under guardianship or subject deprived of liberty
* Opposition to participation in the study

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: University students, teenagers and parents of teenagers to test understanding of linguistic validation of questionnaires
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
The process of validation will be performed by the forward/backward method (Epstein et al. 2015). The translation will be considered valid when the tests performed by the participants are considered successful. | through questionnaires completion, an average of 1 day

SECONDARY OUTCOMES:
Evaluation of the internal consistency of the questionnaires after cross-cultural adaptation in French language | through questionnaires completion, an average of 1 day

IPD SHARING:
Plan to Share IPD: No